CLINICAL TRIAL: NCT02135120
Title: Do Peripheral Nerve Blocks When Used as Part of a Multimodal Regimen Inclusive on Intrathecal Morphine Improve Analgesia After Unilateral Total Knee Arthroplasty? A Randomized Controlled Trial
Brief Title: The Efficacy of Peripheral Nerve Blocks With Intrathecal Morphine in Improving Analgesia After Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ghassan Kanazi, Professor and Chairman, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ANES.GK.09
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia; Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Morphine group (Active Comparator): Patients will receive a combined spinal epidural anesthesia technique with intrathecal morphine
  Interventions: Drug: Combined spinal epidural anesthesia technique with intrathecal morphine
- Morphine-femoral group (Active Comparator): Patients will receive a combination of combined spinal-epidural (with intrathecal morphine) and femoral nerve block
  Interventions: Drug: A combination of combined spinal-epidural (with intrathecal morphine) and femoral nerve block
- Morphine-femoral-sciatic group (Active Comparator): Patients will receive a combination of combined spinal-epidural (with intrathecal morphine) and femoral nerve block as well as sciatic nerve block
  Interventions: Drug: A combination of combined spinal-epidural (with intrathecal morphine) and femoral nerve block as well as sciatic nerve block

INTERVENTIONS:
Drug: Combined spinal epidural anesthesia technique with intrathecal morphine
  Arms: Morphine group
Drug: A combination of combined spinal-epidural (with intrathecal morphine) and femoral nerve block
  Arms: Morphine-femoral group
Drug: A combination of combined spinal-epidural (with intrathecal morphine) and femoral nerve block as well as sciatic nerve block
  Arms: Morphine-femoral-sciatic group

SUMMARY:
The purpose of this study is to determine whether intrathecal morphine (ITM) alone or its combination with peripheral nerve blocks (PNB) provides better analgesia for patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) surgery is associated with severe pain. The success of knee rehabilitation following surgery depends largely on adequate pain control that permits early physical therapy. Postoperative modern analgesic recommendations specific to TKA propose either spinal block with intrathecal morphine (ITM) or a combination of general anesthesia with single shot femoral nerve block (SFNB). Femoral nerve block (FNB) too has proven analgesic advantages in TKA surgery. However, we do not know if the combination of the two analgesic techniques, ITM and peripheral nerve blocks (PNB), provides superior analgesia to ITM alone.

Thus, this study aims to determine whether ITM alone or its combination with PNB provides better analgesia for patients undergoing total knee arthroplasty (TKA).

Eligible patients undergoing unilateral TKA under spinal anesthesia consenting to a multimodal analgesic regimen inclusive of ITM, FNB, and SNB will be recruited. All patients will receive spinal with intrathecal morphine. Patients will be randomly assigned using a computer generated table of random numbers to receive either spinal with intrathecal morphine (morphine group), a combination of intrathecal morphine and femoral nerve block (morphine-femoral group), or a combination of intrathecal morphine and femoral nerve block as well as sciatic nerve block (morphine-femoral-sciatic group).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients undergoing unilateral TKA under spinal anesthesia and nerve blocks
* Ages 18-80
* BMI ≤ 38 kg/m2

Exclusion Criteria:

* BMI > 38 kg/m2
* chronic pain disorders
* Significant pre-existing neurological deficits or peripheral neuropathy affecting the lower extremity
* abuse of drugs or alcohol
* Contraindication to a component of multi-modal analgesia
* Contraindication to spinal anesthesia or failure to institute spinal anesthesia after performing femoral and sciatic blocks
* Bilateral TKA surgeries
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy
* Moderate to severe obstructive sleep apnea.
* Previous adverse reactions resulting from intrathecal opioids (respiratory depression, urinary retention, severe pruritis, severe nausea or vomiting, severe sedation)
* inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Postoperative parenteral morphine consumption | first 24 hours post-operation

SECONDARY OUTCOMES:
Visual analogue pain scores (VAS) in anterior and posterior knee | within 24-48 hours after surgery
Severity of pain in anterior and posterior knee | 1 week postoperatively
Time to first IV PCA bolus | within first 12 hours
Total IV PCA consumption upon discontinuation of PCA | 24-48 hours after surgery
Side effects | within 24 hours after surgery
  Patients will be closely monitored during their hospital stay. Patients will be assessed in their rooms twice daily by a pain nurse, and additionally as required, to report the occurrence of side effects including: block complications, incidence of falls, numbness over femoral distribution, nausea & vomiting, pruritus, occurrence of urinary retention, occurrence of respiratory depression.
Patient satisfaction with pain control | 24-48 hours after surgery
complications | 1 month after surgery
  Patients will be contacted by a member of the research team (by phone) to check for complications including: numbness in the anterior thigh, numbness in the foot, pain and/or bruising around the site where the anesthetic were injected, weakness in thigh muscles, weakness in foot muscles

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan E Kanazi, MD, Principal Investigator — American Univesity of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon